CLINICAL TRIAL: NCT01731080
Title: Arterial Wall Calcium Load and Preferential Sites in Pseudoxanthoma Elasticum Versus Type 2 Diabetes and Chronic Kidney Disease.
Brief Title: Arterial Wall Calcium Load in Pseudoxanthoma Elasticum
Acronym: Ca-Art-PXE2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: AOI-2011
Record Dates: First submitted 2012-11-14; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Pseudoxanthoma Elasticum; Type 2 Diabetes; Chronic Kidney Disease
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Pseudoxanthoma Elasticum: Patients with genetically and clincally proven PXE
- chronic kidney disease: Type 2 diabetic patients with mediacalcosis and matched to PXE patients for gender and age (+/- 5 yrs).
- Diabetes: patients with chronic kidney disease and matched to PXE patients for gender and age (+/- 5 yrs).

SUMMARY:
Quantification and preferential sites of arterial wall calcification within the coronary and lower legs arteries will be comared between Pseudo-Xanthoma elasticum(PXE) atients and type 2 diabetics and Chronic Kidney disease.

DETAILED DESCRIPTION:
In a previous work we have observed that patients suffering from PXE, a soft-tissue calcifying inherited autosomal disease, exhibited specific structural and functionnal features within the peripheral arteries. We now want to quantify and determine the preferential sites of the arterial wall calcification (Agatston score) between these patients compared to diabetics and patients with chronic renal insufficiency with mediacalcosis.

All variables will be collected from a cohort of PXE monitored in our PXE Health and Care centre at the university hospital of Angers. Quantification of the arterial wall calcium load will be performed using helicoidal CT-scan. These variables will be compared to the same measurements performed in type 2 diabetic and chronic kidney disease patients paired by age and gender.

ELIGIBILITY:
Inclusion Criteria:

* Patients with phenotypically and genotypically-proven PXE
* Type 2 diabetic patients with mediacalcosis (i.e. Ankle Brachial Index > 1.30)
* Patients with a chronic kidney disease (CKD), before kidney transplantation
* All patients should be affiliated to a Health care system

Exclusion Criteria:

* Patient with unproved PXE
* Patient under the age of 18 yrs
* Patient unwilling to participate to the study
* Pregnant women
* Patient not affiliated to a Health care system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pseudoxanthoma Elasticum (PXE)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
calcification score | after inclusion
  the level of arterial wall calcification determined by a Ct-scan and computed by the Agatston score

SECONDARY OUTCOMES:
site of calcification | after inclusion
  the anatomical site of arterial wall calcification determined by a Ct-scan and computed by the Agatston score

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE CORRE, MD, Principal Investigator — Department of Dermatology, University Hospital of Angers, France
Locations (1):
- University Hospital, Angers, Pays de la Loire Region, France